



# Non-operative treatment of pediatric lateral humeral condyle fractures: a cohort study of 50 patients

# **Clinical Investigation Plan**

File name: Study Protocol - Non-OP treatment of LHCF - H-21017621.pdf

Version and date: Version 3.0, 30 July 2021

# **Principal Coordinating Investigator**

#### **Morten Jon Andersen**

MD

Department of Orthopedic Surgery Copenhagen University Hospital – Herlev and Gentofte, Copenhagen, Denmark

Phone +45 38 68 14 79 Mobile +45 26 14 86 24

E-mail morten.jon.andersen@regionh.dk

#### **Sponsor**

24

25

26

27 28 Department of Orthopedic Surgery and Department of Radiology and Scanning Copenhagen University Hospital Herlev and Gentofte Copenhagen, Denmark The Danish Data Protection Agency ID: P-2020-1197

The Danish National Committee On Health Research Ethics ID: H-21017621

### **Confidentiality statement**

The information provided in this document is strictly confidential and is available for review to investigators, potential investigators and appropriate Ethics Committees (EC). No disclosure should take place without written authorization from the sponsor, except to the extent necessary to obtain informed consent from potential patients.



Protocol ID: H-21017621 Version 3.0, July 30, 2021

# Content

| 20 | CI | inical Investigation Plan | 4 |
|----|------|-----------------------------------------------------|----|
| 30 | U | Inical Investigation Plan | |
| 31 | | Principal Coordinating Investigator | |
| 32 | | Sponsor | |
| 33 | Α Ι. | Confidentiality statement | |
| 34 | | obreviations/glossary | |
| 35 | | efinitions | |
| 36 | 1 | Synopsis | |
| 37 | 2 | | |
| 38 | 3 | General information/responsibilities | |
| 39 | | 3.1 Responsibilities | |
| 40 | 4 | Background and literature review | |
| 41 | | 4.1 Definition and epidemiology | |
| 42 | | 4.2 Diagnosis | |
| 43 | | 4.3 Outcome | |
| 44 | | 4.4 Current status of research in this area | 9 |
| 45 | 5 | Primary and secondary objectives | 11 |
| 46 | | 5.1 Primary objective | 11 |
| 47 | | 5.2 Secondary objective(s) | 11 |
| 48 | | 5.3 Hypothesis | 11 |
| 49 | 6 | Study design | 11 |
| 50 | | 6.1 Study population and patient enrollment | 11 |
| 51 | | 6.2 Study procedures | 13 |
| 52 | | 6.3 Study treatments | 15 |
| 53 | 7 | Definitions of outcome measures and study variables | 18 |
| 54 | | 7.1 Primary outcome | 18 |
| 55 | | 7.2 Secondary outcomes | 19 |
| 56 | 8 | Statistical planning | 21 |
| 57 | | 8.1 Hypotheses | 21 |
| 58 | | 8.2 Sample size considerations | 21 |
| 59 | | 8.3 Statistical analysis | 21 |
| 60 | 9 | Bias | 21 |
| 61 | 10 | Benefits | 22 |
| 62 | 11 | Risk analysis | 22 |
| 63 | | 11.1 Treatment-related risks | 22 |
| 64 | | 11.2 Study disadvantages | 22 |





90

Version 3.0, July 30, 2021

| 65 | 11.3 Study-related risks | 22 |
|----------|-----------------------------------------------------------|----|
| 66 | 11.4 Actions to minimize increased risks | 23 |
| 67 | 12 Informed consent process | 23 |
| 68 | 12.1 Special considerations to consent pediatric patients | 23 |
| 69 | 13 Adverse event reporting | 24 |
| 70 | 14 Data management | 24 |
| 71 | 14.1 Data collection, source data, storage and archiving | 24 |
| 72 | 14.2 Imaging data | 25 |
| 73 | 14.3 Confidentiality | 25 |
| 74 | 15 Regulatory affairs | 25 |
| 75 | 16 Disclosures and economy | 25 |
| 76 | 17 Patient insurance | 25 |
| 77 | 18 Study report and publication policy | 25 |
| 78 | 18.1 Final Study Report | 25 |
| 79 | 18.2 Publication | 26 |
| 80 | 19 Termination criteria | 26 |
| 81 | 19.1 Stopping rules | 26 |
| 82 | 20 Deviations from the Clinical Investigation Plan | 26 |
| 83 | 21 Amendments to the Clinical Investigation Plan | 26 |
| 84 | 22 Time schedule | 27 |
| 85 | 23 Authors | 27 |
| 86 | 24 Reference list | 28 |
| 87 | Appendix 1 - Diagnosis and Treatment Protocol | 31 |
| 88<br>89 | | |





# 91 Abbreviations/glossary

| | giossaiy |
|---|---|
| AE/SAE | Adverse Event(s)/Serious Adverse Event(s) |
| ADE/SADE | Adverse Device Event(s)/Serious Adverse Device Event(s) |
| AO | Arbeitsgemeinschaft für Osteosynthesefragen = Association for the Study of Internal Fixation (ASIF) |
| CIP | Clinical Investigation Plan |
| CRF | Case Report Form |
| CRO | Contract Research Organization = Clinical Research Organization |
| EC | Ethics Committee |
| eCRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |
| FSR | Final Study Report |
| FU(s) | Follow-up(s), eg follow-up visit(s), follow-up procedure(s) |
| GA | General Anesthesia |
| GCP | Good Clinical Practice |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use |
| ISF | Investigator Site File |
| ISO | International Organization for Standardization |
| LHCF | Lateral Humeral Condyle Fracture |
| MeSH | Medical Subject Heading |
| MRI | Magnetic Resonance Imaging |
| PCI | Principal Coordinating Investigator (= Principal Clinical Investigator) |
| PI | Principal Investigator |
| SD | Standard Deviation |
| U(S)ADE | Unanticipated (Serious) Adverse Device Effect |

# 92 93

### **Definitions**

| Deminions | |
|---|---|
| Baseline | Status post injury but pretreatment |
| Enrolled | Patients with written informed consent who commenced treatment within the study |
| Follow-up visit | FU; visit at predefined times after the treatment day |
| Follow-up population | Patients intended to be followed-up (i.e. enrolled population) |
| Injury day | "Day 0"; day of injury |
| Written informed consent | Legally binding signature on the informed consent form (ICF) (i.e. the patient's parents or legal guardians) |



# 1 Synopsis

| Official title | Non-operative treatment of pediatric lateral humeral condyle fractures: a cohort study of 50 patients |
|---|---|
| Short title | Non-operative treatment of pediatric lateral humeral condyle fractures |
| Sponsor | Department of Orthopedic Surgery<br>Copenhagen University Hospital – Herlev and Gentofte |
| Registration | The study will be registered with ClinicalTrials.gov |
| Background and purpose | The diagnosis of LHCF is complicated by radiographic inability to show the full extent of the injury into the chondral (unossified) epiphysis. MRI gives a perfect view of these fractures. The safety and feasibility of non-operative treatment based on MRI findings in children with elbow fractures has not been investigated in a Danish setting. If safe and feasible, the use of MRI could dramatically lower the need for surgery in children with LHCF. |
| Condition | Pediatric lateral humeral condyle fracture |
| Intervention/procedure investigated | Non-operative treatment of LHCF based on MRI findings |
| Comparison | None |
| Study type | Interventional |
| Study design | Prospective, Cohort, Single center |
| Short description | Cohort study of 50 patients aged 2-15 with acute LHCF. Intervention with non-operative treatment based on MRI performed without sedation or anesthesia. Objectives are to describe functional outcome, radiological healing, secondary fracture displacement and any complications after two years. Patients are seen for follow-up 1, 2 and 4 weeks and 3, 6, 12 and 24 months after injury. The investigators hypothesize that undisplaced and minimally displaced LHCF can be treated non-operatively based on MRI findings with good functional outcomes after two years. |
| Primary objective | Describe the functional outcome two years after non-operative treatment of undisplaced and minimally displaced LHCF in children. |
| Secondary objectives | <ul> <li>Describe the feasibility of performing a subacute MRI of the elbow in children with LHCF within 2-7 days after the injury without sedation or anesthesia</li> <li>Report MRI findings and classify fractures according to Song classification based on MRI</li> <li>Report the number and proportion of fractures that displace secondarily and their treatment</li> <li>Report final treatment; non-operative or operative</li> <li>Describe radiographic results and compare with MRI</li> <li>Report any early or late complications</li> </ul> |



Hypothesis Children with minimally displaced LHCF (Song stage 1, 2 and 3) can be treated non-operatively based on MRI findings with good functional outcome after two years. Primary outcome Mayo Elbow Performance Score (MEPS) two years after injury measure Secondary outcome Pain measures Radiographic results MRI results Alteration in treatment regime based on MRI Number and proportion of fractures with secondary displacement Any early or late complications Statistical Sample size is estimated from previous studies which included less than considerations and 30 participants. The investigators of this study suspect that by enrolling estimated enrollment 50 participants the age distribution and variation in fracture pattern will be representative of the background population. Baseline characteristics and outcomes recorded at scheduled FU assessments will be presented using simple summary statistics. Start of enrollment October 2021 (estimated) Last patient/last visit October 2025 (estimated) Eligibility inclusion Inclusion criteria: criteria Children age 2-15 years Diagnosis of acute LHCF (<5 days) with <5 mm of displacement on plain radiographs Parental informed consent obtained Eligibility exclusion Exclusion criteria: criteria Contraindication(s) to performing an MRI Unable to participate in follow-up Existing bone pathology Previous ipsilateral elbow fracture **Principal Coordinating** Morten Jon Andersen, MD Investigator Department of Orthopedic Surgery Copenhagen University Hospital – Herlev and Gentofte Copenhagen, Denmark Phone +45 38 68 14 79 Mobile +45 26 14 86 24 E-Mail morten.jon.andersen@regionh.dk Study site Department of Orthopedic Surgery Copenhagen University Hospital – Herlev and Gentofte Copenhagen, Denmark Health authority The Danish Data Protection Agency The Danish National Committee On Health Research Ethics



Non-operative treatment of pediatric lateral humeral condyle fractures


| Pubmed Medical<br>Subject Heading<br>[MeSH] terms and<br>keywords | Child [MeSH] Casts, Surgical [MeSH] Fracture Fixation [MeSH] Humeral Fractures [MeSH] |
|---|---|
| Imaging review | All images collected will be analyzed by independent radiologists during the study |

96



98

109

115

Non-operative treatment of pediatric lateral humeral condyle fractures


# 2 Rationale and purpose of the study

The treatment of LHCF is most often surgical with open reduction and fixation [1]. The diagnosis of 99 LHCF is complicated by radiographic inability to show the full extent of the injury into the unossified 100 chondral epiphysis and therefore physicians often opt for open surgical treatment. MRI; however, gives 101 a perfect view of these fractures [2-5]. This project investigates the safety and feasibility of non-102 operative treatment of LHCF based on MRI performed without sedation or anesthesia and seeks to 103 dramatically lower the need for surgery. Objectives are to describe functional outcome, radiological 104 healing, secondary fracture displacement and any complications after two years. The investigators 105 hypothesize that undisplaced and minimally displaced LHCF can be treated non-operatively based on 106 MRI findings with good functional outcomes after two years. A cohort study design is used to follow 50 107 children with LHCF. 108

# 3 General information/responsibilities

- The International Conference on Harmonization for Good Clinical Practice (ICH-GCP) and ISO 14155 guidelines define the responsibilities of the sponsor and investigators in the context of the study. Specific topics, such as the permission from the responsible EC, are defined separately in the CIP. The study site undertakes to guarantee correct and prompt implementation, documentation, and transmission of the study data.
- In the context of the study, the participating study site will return the completely documented cases.

  Completely documented means that all FU visits have been carried out for the cases included in the

  study and that these assessments are recorded on the electronic Case Report Forms (eCRFs) specially

  designed for this study. Furthermore, the necessary radiological investigations must be performed at the

  FU visits.

#### 121 3.1 Responsibilities

### Principal Coordinating Investigator Morten Jon Andersen MD

Department of Orthopedic Surgery Copenhagen University Hospital - Herlev and Gentofte, Copenhagen, Denmark

Phone +45 38 68 14 79 Mobile +45 26 14 86 24

E-Mail morten.jon.andersen@regionh.dk

### Sponsor Copenhagen University Hospital Herlev and Gentofte

Department of Orthopedic Surgery and Department of Radiology and Scanning Copenhagen University Hospital Herlev and Gentofte Copenhagen, Denmark

122

123

124 125







# 4 Background and literature review

| | | | | _ |
|-----|------------|--------|-------|-------|
| 4.1 | Definition | and en | idemi | oloav |

128129130

131

132

127

Fractures of the distal humerus account for 5-10% of all pediatric fractures but constitute up to 30% in children aged 4-9 years of age [6–10]. Fractures of the lateral humeral condyle account for 10-20% of all elbow fractures in children making it the second most frequent after supracondylar fractures [3,11,12].

133134135

136

137

LHCF are usually the result of a fall on an outstretched arm with either the extensor-supinator mass pulling or the radial head pushing off the lateral condyle [13]. The diagnosis is suspected by the history of a fall, usually a swollen and painful elbow with tenderness over the lateral aspect. In more severe cases a hematoma can present early.

138139140

141

A LHCF is a Salter-Harris type II or IV physeal fracture which can appear as everything from a hairline fracture to grossly displaced intraarticular injuries.

#### 4.2 Diagnosis

142143144

145

146

147

149

150

Fractures are usually diagnosed on plain radiographs with antero-posterior (AP), medial-lateral (ML) and internal oblique (IO) radiographs. Especially the IO is important in appreciating the amount of displacement [14]. The distal humerus, especially in younger children, is largely composed of cartilage and is termed the chondroepiphysis [7]. Four secondary ossification centers arise with growth at different ages making interpretation of elbow radiographs in children a challenge [15]. A study showed that emergency department (ED) physicians only made the right radiographic diagnosis in 53% (16/30) of cases concerning pediatric elbow injuries [16].

151 152

#### 4.3 Outcome

Neglecting to treat displaced LHCF can lead to painful nonunion, malunion and growth disturbances e.g. fishtail deformity. Complications such as tardy ulnar nerve palsy and varus or valgus deformity can

develop years after an untreated injury [13].

#### 4.4 Current status of research in this area

156157158

159

160

Undisplaced and minimally displaced LHCF found on radiographs compose a specific challenge in choosing between non-operative or operative treatment [13]. The risk of secondary displacement of an initially undisplaced fracture varies from 4% to more than 40% depending on the initial stability and displacement [12].

161162163

Historically these fractures where classified according to Milch [17] however this system neither describes fracture stability nor focusses on fractures in children and has no prognostic value [1].

164165166

Song's classification (figure 1) [18] discerns incomplete from complete and undisplaced from displaced fractures clearly describing fracture stability.

167168

Song stage 1 fractures only involve the bony metaphysis. Stage 2 fractures pass into the chondroepiphysis, but not through, leaving the articular cartilage intact and functioning as a hinge [4].







Figure 1 - Song classification.

Because of the risk of secondary displacement, operative treatment is often conducted with many surgeons choosing open reduction and fixation in all cases [19,20]. Operative fixation imposes the risk of minor complications such as superficial infection, ulcers and granulomas but also major complications such as deep infection, osteomyelitis, malunion, non-union, growth disturbance and osteonecrosis [21].

MRI with specific cartilage sequences (figure 2) can clearly show the chondroepiphysis and studies have shown that MRI is capable of precisely showing the fracture pattern [2,3,5,22]. Using simple techniques and advances in technology to prepare the child, MRI has been shown to be feasible in younger children without sedation or anesthesia in whom this was previously thought necessary [23–30].



Figure 2 - MRI showing LHCF. Left: Stage 1, confined to metaphysis. Center: Stage 2, fracture line stops in the chondroepiphysis. Right: Stage 3, traverses the joint cartilage.





# Primary and secondary objectives

| 197 | 5.1 | Primary of | objective |
|-----|-----|------------|-----------|
|-----|-----|------------|-----------|

198 199

200

196

To describe the functional outcome two years after non-operative treatment of undisplaced and minimally displaced LHCF in children.

#### 5.2 Secondary objective(s) 201

202 203

204

- Describe the feasibility of performing a subacute MRI of the elbow in children with LHCF within 2-7 days after the injury without sedation or anesthesia
- Report MRI findings and classify fractures according to Song classification based on MRI 205
- Report the number and proportion of fractures that displace secondarily and their treatment 206
- Report final treatment; non-operative or operative 207
- Describe radiographic results and compare with MRI 208
- · Report any early or late complications 209

**Hypothesis** 

#### 210 211

5.3

Children with minimally displaced LHCF (Song stage 1, 2 and 3) can be treated non-operatively based 212 on MRI findings with good functional outcome after two years. 213

#### Study design 214

- This project uses a cohort study design conformed to the STROBE Statement [31]. The investigators 215
- aim to prospectively and consecutively recruit all children with undisplaced or minimally displaced LHCF 216
- (cohort) which based on MRI are treated non-operatively (exposure). We report functional and 217
- radiological outcome two years after the injury (outcome). This study design is relevant in reporting the 218
- primary and secondary outcomes based on the exposure in our cohort. 219

#### 6.1 Study population and patient enrollment

220 221

This study investigates the treatment of pediatric LHCF; therefore, this study cannot be conducted in 222 consenting adults. LHCF occur predominantly in 4-9 year olds and thus it is not possible to select only 223

older children for inclusion. 224

225 226

227

This study is believed to have great positive implications for the participants and successive patients with the same condition.

#### 6.1.1 Setting 228

- The study will be performed in the Capitol Region of Denmark. Patients in the catchment area of 229
- Copenhagen University Hospital Herlev and Gentofte are eligible for recruitment (population 700.000 230 of which 80.000 are children).
- 231



Non-operative treatment of pediatric lateral humeral condyle fractures Protocol ID: H-21017621

Version 3.0, July 30, 2021

| 233 | 6.1.2 | Inclusion | criteria |
|-----|-------|-----------|----------|

- Children aged 2-13 years 234
- Diagnosis of acute LHCF 235
- Fracture <5 days old</li> 236
- Fracture with <5 mm of displacement on plain radiographs (AP, ML and IO views)</li> 237

238

240

- Parental informed consent obtained: 239
  - Ability of all legal guardians to understand the content of the patient information and ICF
- Willingness and ability to let the child participate in the clinical investigation according to the 241 Clinical Investigation Plan (CIP) 242
- Signed and dated EC-approved written parental informed consent sheet 243

#### 244 6.1.3 Exclusion criteria

- Contraindication(s) to performing an MRI [32] without the use of sedation or anesthesia: 245
- Ferromagnetic implants or foreign bodies 246
- Pacemaker 247
- Ear implant 248
- Severe claustrophobia 249
- · Unable to participate in follow-up 250
- Existing bone pathology 251
- Tumor 252
- Osteogenesis imperfecta 253
- Degenerative disease 254
- Previous ipsilateral elbow fracture 255

#### **Enrollment of participants** 256

A member of the research team will identify all eligible patients (i.e., who meet all of the inclusion and none of the exclusion criteria).

258 259 260

257

The identification of eligible patients is done during the daily routine review of radiographs taken in the ED of Copenhagen University Hospital - Herlev and Gentofte.

261 262 263

264

265

266

267

Electronic letters for FU cannot be sent to minors; therefore all parents are routinely approached by phone. During this standard approach we ask permission from the EC to inquire the parents about their interest and their child's eligibility in participating in this study. This inquiry will include a short prescreening with questions to confirm eligibility as well as a short description of the study and responsibilities for participating. None of the data of the pre-screening process will be documented study specifically.

268 269 270

271

272

If interested in participating, the parents and the patient are invited to the outpatient clinic. Parents are informed of the possibility of bringing an assessor. At the visit, a member of the research team will go through the informed consent process, and explain the purpose of the study, the procedures, the risk/benefits, alternatives to participation, and data protection.

273 274 275

276 277 For each patient participating the parents will sign and date an ICF. A copy of the signed ICF will be placed into the ISF and one copy will be handed over to the parents. A more detailed description of the informed consent process is provided in section 12.







All patients with written informed consent will be allocated to a unique patient trial number. The date of informed consent and the recruitment information is entered in the study database.

279280281

278

The recruitment period will be up to 24 months, during which 50 patients are planned to be enrolled.

# 6.2 Study procedures

282 283 284

285

The schedule of all FU visits including imaging procedures as well as the data to be collected at each visit is shown in Table 1. All FU visits with the defined time windows are calculated from the day of injury (i.e. day 0).

286287288

289

290291

292

All participants live in the catchment area of Herlev and Gentofte Hospital within short transportation time. Information about the time and place for the follow-up examination is sent physically by mail to the current address registered in the Civil Registration System and via the electronic health record (EHR) system. Parents are usually very keen to take their children for follow-up appointments making the risk of missing an appointment low. Any participants who miss an appointment will be contacted by phone to reschedule.

293 294

Table 1: Study schedule

| 295 |
|-----|
| 296 |

| Assessment parameters | Out-patient clinic visits and imaging procedures * | | | | | | | res * | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Visit<br>1** | Visit<br>2 | Visit<br>3 | Visit<br>4 | Visit<br>5 | Visit<br>6 | Visit<br>7 | Visit<br>8 | Visit<br>9 | Visit<br>10 |
| | Injury (day 0) | Screening | Information visit | Enrollment and consent | 5 (± 3) days | 12 (± 3) days | 4 weeks | 3 months | 6 months | 12 months | 24 months |
| Eligibility | | Х | | | | | | | | | |
| Patient information | | | Х | | | | | | | | |
| Consent | | | | Х | | | | | | | |
| Demographics | | | | X | | | | | | | |
| MRI | | | | | Х | | | | | | |
| If applicable - Control-MRI | | | | | | (X) | | | | | |
| Cast removal*** | | | | | | | Х | | | | |
| Radiographs and clinical exam | | | | | | X | X | X | X | X | Х |

297298

300 301

<sup>\*</sup> All FU visits with the defined time windows are calculated from the day of injury (i.e. day 0).

<sup>\*\*</sup> Telephone interview.

<sup>\*\*\*</sup> Casting may be prolonged two weeks in case of lack of callus formation at four weeks.





| 302 <b>6.2</b> | 2.1 Visit | : 1: S | creenin | g (by | phone) |
|----------------|-----------|--------|---------|-------|--------|
|----------------|-----------|--------|---------|-------|--------|

As described in section 6.1.4, the parents of potential study patients are informed about the study 303 over telephone by the PI. 304

#### 6.2.2 **Visit 2: Information visit** 305

- All inclusion and exclusion criteria are checked to decide if the patient can participate in the study.
- Specific procedures for enrollment of pediatric patients are undertaken. A more detailed description 307 of the enrolment of participants and informed consent process is provided in section 6.1.4 and 10. 308
- · Before any study-specific examinations are performed, the patient's parents give written informed 309 consent to participate in the study according to the CIP. 310

#### Visit 3: Enrolment, consent and preparation for MRI 311

- Obtain baseline demographics 312
- Book MRI 313

306

- Prepare child for MRI using the Child Centered Care model described in section 6.3 314
- · Data verification and entry into the eCRF 315

#### 6.2.4 Visit 4: MRI (5 (± 3) days) 316

- The MRI is performed according to the Child Centered Care model described in section 6.3 317
- Results of the MRI are given to the parents by phone 318
- Any necessary adjustments to the treatment plan is made 319
- Entry into the eCRF 320

#### ONLY if applicable: Control-MRI (12 (± 3) days) 6.2.5 321

- If an unstable Song stage 3 fracture is diagnosed based on the initial MRI an additional control MRI 322 is performed during this visit 323
- Results of the MRI are given to the parents by phone 324
- Any necessary adjustments to the treatment plan is made 325
- Entry into the eCRF 326

#### Visit 5: Radiographs and clinical examination (12 (± 3) days) 327

- Plain radiographs of injured elbow without cast (AP, ML and IO)
- Clinical examination 329

328

330

338

- Cast condition
- Assessment of pain and use of pain medication 331
- Neurovascular status of the hand 332
- Entry into the eCRF 333

#### 6.2.7 Visit 6, 7, 8, 9 and 10: Radiographs and clinical examination (4 weeks and 3, 6, 12 and 24 334 months). 335

- Plain radiographs of injured elbow without cast (AP, ML and IO) 336
- Clinical examination 337
  - Assessment of pain and use of pain medication
- Neurovascular status of the hand 339
- Bilateral elbow assessment according to Mayo Elbow Performance Score (MEPS) 340
- Bilateral carrying angle of the elbow measured in degrees by goniometer 341
- · Entry into the eCRF 342



Non-operative treatment of pediatric lateral humeral condyle fractures


| 343 | 6.2.8 | Unscheduled | visits |
|-----|-------|-------------|--------|
|-----|-------|-------------|--------|

- Unscheduled visits can take place at any time during the study if a need occurs or if the investigator
- considers this to be appropriate for patient care. Information collected between study visits are to be
- documented at the next regular study visit with the following exceptions:
- If a patient drops out of the study, a dropout form is completed at the time of dropout

#### 348 6.2.9 Premature study termination

- Patient participation in the study may end prematurely for one of the following reasons:
- Patient withdrew informed consent
- Protocol violation
  - Investigator's discretion (e.g. patient noncompliance with CIP)
- Unknown/lost to FU

354 355

352

For each case of premature termination detailed information will be obtained explaining the circumstances leading to the termination. This will be recorded on a dropout form in the eCRF.

356 357 358

359

- If patients are withdrawn from the study, any collected data will be censored. Censoring allows this collection of data to be accounted for in the analysis.
- 6.3 Study treatments

360 361

364

This study is not investigating any medical device. All devices in this study will be used per standard of care at the participating institutions.

#### 6.3.1 Emergency treatment

- All patients who sustain a LHCF are initially treated in the ED with an above elbow splint. Parents and,
- when applicable, the patient are informed of the injury, cast management and use of pain medicine.

#### 367 6.3.2 MRI in children without sedation or anesthesia

- Child Centered Care (CCC) (figure 3 and 4) consists of:
- Oral and written information about MRI together with a demonstration of the process using a toy scanner is given by a member of the research team to parents and patient.
- Movies from the hospital's radiology department that prepare the child for the experience.
- An interactive app (Rumble in MRI, free in App Store and Google Play Store) that prepares and motivates the child. The troll character Rumble and 3D animations of rooms increase recognisability.
  - A pediatric team of radiographers focus on the child feeling safe and secure.
    - A child-friendly environment in the MRI room with lights and movies coordinated in themes known from the app projected on the wall ("Philips Ambient Experience", Philips Electronics, Koninklijke, Netherlands).

377378

374

375





Figure 3 - Left) Rumble in MRI app. Right) Toy scanner from Playmobil® used to show children the procedure.

To further better the child's experience, all MRIs are performed during daytime hours, preferably before noon. Parents are asked to give the child pain medicine according to age and weight before leaving home. Scans are performed with an above elbow splint on.

### 6.3.3 MRI protocol

MRI examination (figure 4) of the elbow is performed using Philips dStream S flex coils on 3 Tesla MRI scanners (Philips Ingenia Elition X 3T and Philips Ingenia 3T). Patients undergoing the examination will have a splint on with the elbow flexed to 90 degrees. The splinted elbow is lowered beside the patient, removing the respiratory artifact. The dStream S flex coils include two flexible coils which can obtain 10 cm coverage with a maximum of four channels. These coils are placed around the patients elbow parallel to each other, and perpendicular to the static magnetization field.







Figure 4 – A pediatric team of radiographers focus on the child feeling safe and secure.

The MRI protocol consists of three sequences with breaks in between; 3D WATS - 2 minutes and 32 seconds, T1 coronal – 2 minutes and 16 seconds and STIR coronal 3 minutes and 53 seconds. Total scan time is less than 9 minutes. The most important information comes from the 3D WATS sequence and in most cases the derived images will be sufficient to choose between non-operative or operative treatment.

In total, 45 minutes is set aside for receiving and briefing patient and parents, positioning the child and completing the scans. Parents are invited to sit next to the child during the scan. The radiographers involve the children by dialog and each child can choose the color of the room. The child holds the stop







button in his or her hand, so that they can press stop along the way. Communication with radiographers is possible throughout the procedure. The procedure is stopped at any request from the child or parents or if deemed necessary by the radiographers.

407 408 409

410

411

412

413

405

406

#### 3D Water Selective Excitation (WATS)

3D WATS is a fast field echo T1 weighted pulse sequence [33]. 3D WATS utilizes the chemical shift artifact to differentiate between the frequencies of fat and water. The sequence applies a technique where the water protons are selectively excited to induce fat suppression in cartilage. WATS is a 3D imagery so it can be reconstructed with various slices in the computer after the scan. The 3D WATS sequence is usually used for evaluation of cartilage.

414 415 416

417

418

#### T1

T1 weighted images results from the differences in the T1 recovery times of the tissues. In T1 sequences, fat and degeneration has a high signal, where cortical bone, infection and cysts has a low signal. T1 weighted images are used to portray the anatomy.

419 420 421

422

423

### **Short Tau Inversion Recovery (STIR)**

STIR is a pulse sequence that suppresses the signal from fat [34]. STIR is an important sequence in musculoskeletal imaging showing lesions inside of the bone. A normal bone contains fat bone marrow and STIR suppresses fat which shows lesions with bone marrow edema.

424 425 426

427

431

Table 2: Specific scan parameters and scan times

| Parameter | 3D WATS | T1 COR | STIR COR |
|---|---|---|---|
| TR | 20 | Range (450-750) 750 | 3536 |
| TE | 4.9 | 9 | 60 |
| FA | 15 | 90 | Inversion Recovery: 220 msek. |
| | | | Refocusing angle: 90* |
| Scan mode | 3D | 2D | 2D |
| Technique | FFE | SE (TSE) | IR (TSE) |
| Slice thickness | 3 mm | 3 mm | 3 mm |
| Interslice gap | -1.5 mm | 0.3 mm | 0.3 mm |
| FOV | 150 x 150 | 140 x 140 | 130 x 130 |
| Voxel | 0.493 x 0.493 | 0.5 x 0.53 | 0.6 x 0.74 |
| Time | 2.32 min | 2.16 min | 3.53 min |

#### 6.3.4 MRI results

- The results of the MRI are reconstructed and read by senior MRI radiologists together with the PI.
- Patient and parents are informed of the MRI findings and the following treatment (operative or non-
- operative) by the PI.

#### 6.3.5 Operative treatment

- 432 If the MRI cannot be completed for any reason, the images are insufficient in establishing fracture
- pattern or if the MRI shows an unstable fracture which is displaced more than 2 mm, we will suggest
- operative treatment with Kirschner wire fixation. Further participation in this project will be terminated.







#### 6.3.6 Non-operative treatment

Patients with undisplaced and minimally displaced LHCF as seen on MRI will follow a non-operative treatment protocol (appendix 1). The treatment consists of an above elbow splint until radiographic union. Radiographic union usually occurs after four weeks; however, treatment will be continued until callus formation is seen at the cortex of the metaphysis.

Fractures that are not complete (e.g., do not traverse both metaphysis, physis, epiphysis and joint cartilage) are considered stable. Complete fractures displaced <2 mm are considered unstable but still eligible for non-operative treatment. All patients will be seen for FU as outlined in section 6.2.

Any patient with a fracture seen to displace more than 2 mm during FU will be suggested operative treatment.

# 7 Definitions of outcome measures and study variables

### 7.1 Primary outcome

#### 7.1.1 Mayo Elbow Performance Score (MEPS)

MEPS consists of four domains; pain, elbow range of motion (ROM), stability and function [35]. We use a modified MEPS which omits the functional domain because it is not relevant in smaller children. The total score ranges from 0-100 with higher scores indicating better function (figure 5). If the total score ranges between 75 and 100, the result is good (satisfactory); 50–74, fair (acceptable); <50, poor (unsatisfactory) [36]. MEPS has been found to be accurate and reliable compared to other elbow scoring systems [37].

| Criteria | No. of |
|-------------------------------------------|--------|
| | points |
| PAIN (max., 60 points) | |
| None | 60 |
| Mild to occasional, no medication | 40 |
| Moderate to occasional, activity limited, | 20 |
| medication | |
| Severe to incapacitating | 0 |
| MOTION (max. 30 points) | |
| Arc of extension/flexion: | |
| >90 | 30 |
| 60–89 | 20 |
| 30-59 | 10 |
| <30 | 0 |
| STABILITY (max., 10 points) | |
| Effect on function of the elbow | |
| None or mild (does not limit activity) | 10 |
| Moderate (impairs certain functions) | 5 |
| Severe (markedly limits activity) | 0 |

Figure 5 - Modified Mayo Elbow Performance Score.



Non-operative treatment of pediatric lateral humeral condyle fractures


#### 7.2 Secondary outcomes

#### 460 **7.2.1 MRI results**

- Proportion of successful MRIs defined as a completed scan with an image quality that is useful for analysis by the radiologist.
- MRI findings.

459

- Song classification based on MRI.
- Scan length (minutes).
- Any discomforts for the child during the scan.

#### 467 **7.2.2 Radiographic results**

- Injury radiographs and subsequent radiographs during FU will be read and described by a senior
- orthopedic surgeon.

#### **7.2.3 Secondary displacement**

- Any secondary displacement and amount of radiographic displacement (mm) is recorded.
- 472 **7.2.4 Pain**
- To quantify pain in the patient, an age appropriate rating scale is applied:
- Age <5 years: Face, Legs, Activity, Cry, Consolability Scale (FLACC)</li>
- Age >4 years: Faces Pain Scale Revised (FPS-R)
- Age >8 years: Visual analogue scale

477 478

479

480

#### Face, Legs, Activity, Cry, Consolability Scale (FLACC)

To quantify pain behaviors in children who may not be able to verbalize the presence or severity of pain FLACC [38] provides a simple framework. The child is observed for at least 2-5 minutes. Legs and body are observed uncovered. Activity is observed and body is assessed for tenseness and tone.

| 481 |
|-----|
| 482 |

| Behavior | 0 | 1 | 2 |
|---|---|---|---|
| Face | No particular expression or smile | Occasional grimace or frown, withdrawn, disinterested | Frequent to constant quivering chin, clenched jow |
| Legs | Normal position or relaxed | Uneasy, restless, tense | Kicking or legs drawn up |
| Activity | Lying quietly, normal position, moves easily | Squirming, shifting, back and forth, tense | Arched, rigid or jerking |
| Cry | No cry (awake or asleep) | Moans or whimpers; occasional complaint | Crying steadily, screams, sobs, frequent complaints |
| Consolability | Content, relaxed | Reassured by touching, hugging or being talked to, distractible | Difficult to console or comfort |

483 484

485

486

487

Assessment of Behavioural Score:

- 0 = Relaxed and comfortable
- 1-3 = Mild discomfort
  - 4-6 = Moderate pain
- 7-10 = Severe discomfort/pain

489

490

491

492

AO Foundation | AO Education Institute Stettbachstrasse 6 | 8600 Duebendorf | Switzerland Phone: +41 81 414 21 11 | E-mail: aopeer@aofoundation.org | www.aopeer.org







### Faces Pain Scale - Revised (FPS-R)

The Faces Pain Scale – Revised (FPS-R) [39] is used to quantify pain in children above four years of age. It is a self-report measure of pain intensity developed for children. It was adapted from the Faces Pain Scale [40] to make it possible to score the sensation of pain on a 0-to-10 metric. The scale shows a close linear relationship with visual analog pain scales (VAS) across the age range of 4-16 years.













499 500

493

494

495

496

497 498

Figure 6 - Faces of the FPS-R. The child is instructed to point to the faces that shows how much pain the child is in at that moment. Faces are scored 0, 2, 4, 6, 8 or 10 from left to right.

502 503

504

501

FPS-R is easy to administer and requires no equipment except for the photocopied faces (figure 6). The child is asked to point to the face that shows how much pain the child is in at that moment. Faces are scored 0-10 so 0 equals no pain and 10 equals very much pain.

505 506 507

#### Visual analogue scale

508 509

510

511 512

513 514

A visual analogue scale (VAS) (Figure 7) is used to quantify pain in children age 8 and above. VAS has been extensively investigated in quantifying pain in older children [41,42]. The child is asked to put a mark on the line corresponding to the child's pain at that moment. A mark to the far left equals no pain and a mark to the far right equals worst possible pain. The line is 10 cm long and the child's mark is measured from left to right in cm with one decimal e.g., 3.4 cm equaling a VAS of 3.4. If the child cannot cooperate to using VAS, FPS-R is used instead.

515



516

Figure 7 - Visual analogue scale (VAS) for quantifying pain in children age 8 and above.

519 520

518

521





# Statistical planning

| 8.1 Hv | potheses |
|--------|----------|
|--------|----------|

524 525

523

- Minimally displaced LHCF (Song stage 1, 2 and 3) can be treated non-operatively based on MRI 526 findings with good functional outcomes after two years. 527
- 8.2 Sample size considerations 528

529

- Samples size is estimated from previous studies which included less than 30 participants [22,23]. The 530 investigators of this study suspect that by enrolling 50 participants the age distribution and fracture 531 pattern variation will be representative of the background population. By enrolling 50 patients the 532 investigators suspect that any frequent and serious complications will be found. 533
  - Statistical analysis 8.3

534 535

Baseline characteristics and outcomes recorded at scheduled FU assessments will be presented using 536 simple summary statistics. 537

538 539

540

541

- Categorical variables will be summarized using the frequency and percentage for each category.
- Continuous variables will be summarized using the mean, standard deviation (SD), median, interquartile range, and minimum and maximum values and, if appropriate, according to clinically relevant categories.

542 543 544

In general, continuous variables with both baseline and FU measurements available will also be summarized in terms of the individual patient-level changes between baseline and follow-up.

545 546 547

548

554

A p-value of <0.05 is regarded as being significant. Data will be analyzed using SPSS (SPSS, Chicago, IL, USA).

#### 8.3.1 **Patient discontinuation** 549

- If a participant chooses to discontinue the follow-up examinations for any reason, the date and reason 550 for drop-out is recorded and the latest examination will be carried forward in the analysis. In case of 551 drop-out before the first follow-up visit the participant will be excluded from the analysis. Participants are 552 only removed from the study if they decline participation. 553
  - 9 Bias
- We strive to minimize bias in our study. Minimally displaced fractures of the elbow can go unnoticed and 555 be missed by our project. However, Danish parents are usually not withholding in taking an injured child 556 to the ED. A strict protocol for referrals for treatment are in place in Denmark. All eligible patients 557 referred to Herley and Gentofte University Hospital will be asked to participate in the study. We 558 speculate that by enrolling 50 participants the cohort will be representative of the background 559 population. We speculate that these efforts will limit selection bias. Efforts described in the follow-up 560 section reduce the risk of loss to follow-up. Overall, we find a low risk of bias in our study for the chosen 561 study design and size. 562



Non-operative treatment of pediatric lateral humeral condyle fractures


| 1 | n | Bal | nefite | |
|---|---|-----|--------|---|
| 1 | u | Del | nems | ÷ |

Classifying lateral condyle fractures and establishing whether they are stable or not is the key to choosing the right treatment strategy. MRI is the only feasible image modality that can make that distinction.

567 568

569

570

563

LHCF is currently a fracture that requires open surgery in most cases due to the radiographic inability to distinguish stable injuries from unstable. This project seeks to use MRI without sedation or GA in order to distinguish fracture patterns. MRI has been shown to be feasible in all age groups without the need for sedation or GA [24].

571572573

574

575

Thévenin-Lemoine et.al. found that 25 of 27 children could successfully complete an MRI without sedation or GA [23]. Of the 25 children, 17 (68%) had incomplete stable fracture patterns and six (24%) had complete but minimally displaced fractures. In all, 23 (92%) children could be treated non-operatively. Two children had unstable and displaced fractures and underwent surgery.

576577578

If proven safe and feasible, non-operative treatment for undisplaced and minimally displaced LHCF would relieve the child of hospital admission, anesthesia and surgery and reduce parent's need for time off work and reduce overall healthcare costs.

580 581 582

583

584

593

596

597

579

The investigators suspect a significant decrease in the need for operative management based on the results of this project.

### 11 Risk analysis

The risks that occur in this study are associated with the general risks of non-operative treatment for LHCF.

### 587 11.1 Treatment-related risks

- 588 Discomforts/risks from casting:
- Heat injury
- Pressure sores and skin breakdown
- Dermatitis
- Joint stiffness

#### 11.2 Study disadvantages

Extra visits to the outpatient clinic. We follow all patients with seven visits to the outpatient clinic. This is four more than with standard treatment and might be viewed as a disadvantage.

#### 11.3 Study-related risks

#### 11.3.1 Secondary displacement

- During non-operative treatment of fractures, the risk of secondary displacement is well known. The risk
- of secondary displacement of an initially undisplaced LHCF varies from 4% to more than 40%
- depending on the initial stability and displacement [12]. As the initial stability in this study is evaluated by
- 601 MRI the investigators suspect that the risk of secondary displacement will be close to 4%.



Non-operative treatment of pediatric lateral humeral condyle fractures


| 602 | 11.3.2 Radiation | |
|-----|--------------------------|----|
| 603 | In comparison with the s | ta |

In comparison with the standard follow up of LHCF there are four additional visits to the out-patient clinic

- with radiographs of the elbow in AP, ML and IO view. Collectively, the effective dosage is 0.004 mSv -
- far below 0.1 mSv and is considered insignificant.

#### 606 **11.3.3 Loss of privacy**

Patients' private and confidential medical information may get disclosed and confidentiality broken.

607 608 609

#### 11.4 Actions to minimize increased risks

General treatment-related risks will be present whether the patient participates in the study or not. Such risks will be managed by use of standards of treatment, i.e. casting by trained physicians and nurses.

611612613

610

Risk of unnoticed secondary displacement is lowered by an increased number of FUs with radiographs and MRI in case of unstable injury.

614 615 616

The risk of loss of privacy and confidentiality will be managed by strict adherence to data safety and security procedures explained elsewhere in this CIP.

617 618

622

623

624

625

The study will be implemented according to current valid international guidelines (ICH-GCP and ISO

620 14155). The ethical position is based on the Declaration of Helsinki, thus guaranteeing optimal

protection of patient interests.

# 12 Informed consent process

#### 12.1 Special considerations to consent pediatric patients

In this pediatric study, the parent(s) or legal guardian(s) are informed face-to-face about the study and provide informed consent using specific patient information and ICF. In any case, the child is informed orally in an adequate way.

626627628

Written informed consent needs to be obtained from the parent(s) or legal guardian(s). Assent is obtained from any child considered to be able to understand the basic information provided.

629 630

632

633

A member of the research team will, in an undisturbed environment, explain using a plain,

understandable language, movies and toys to each participant and parents the nature of the study, its

purpose, the procedures involved, the expected duration, the potential risks and benefits and any

discomfort it may entail.

635 636

Parents and children will be informed that the participation in the study is completely voluntary and that they may withdraw from the study at any time and that withdrawal of consent will not affect subsequent medical assistance and treatment.

638 639 640

637

The participant's parents will be informed that their child's medical records will be examined directly by authorized individuals involved in the study.

641642643

Consent will be obtained from every patient's parents before any study-specific procedures or assessments take place.



Non-operative treatment of pediatric lateral humeral condyle fractures Protocol ID: H-21017621

Version 3.0, July 30, 2021

| Parents will be provided specific information and ICF describing the study and providing sufficient |
|---|
| information for the parents to make an informed decision about their child's participation in the study |
| together with general information about participating in a research project from the Danish National |
| Committee on Health Research Ethics. |

649650651

646 647 648

Parents will in most cases have at least 24 hours to consider enrollment however, there might be factors (e.g. late presentation to the ED) that dictate more emergent treatment requiring consent with less consideration time.

653654655

656

657

658

659

652

The parents will signify their willingness to let their child participate in the study by signing and dating a personal copy of the approved ICF. The consent form must also be signed and dated by a member of the research team and it will be retained as part of the study records. The investigator will keep the original ICF in the ISF and provide the patient's parents with a copy.

# 13 Adverse event reporting

In this clinical investigation no medical devices are used and based on the risk analyses, AEs or serious
AEs (SAEs) according to ISO 14155 are not collected.

# 14 Data management

This project complies with the EU's General Data Protection Regulation (GDPR) according to the Danish law on data protection *Databeskyttelsesloven* and *Databeskyttelsesforordningen*.

664 665 666

667

668

669

662

663

In order to plan and conduct visits we ask that consent is given to access the patient's EHR. We ask permission to retrieve patient-related data and to read entries regarding visits. We ask permission to access radiographs and MRIs. We ask that access the patient's EHR is given until the conclusion of the project. No access to the patient's EHR regarding the study is made before informed consent to participate is given.

670671672

673

674

675

676

Consent gives the person responsible for the trial and the relevant authorities direct access to obtain information in the patient's medical records for the purpose of carrying out the project as well as for control purposes.

### 14.1 Data collection, source data, storage and archiving

Data management will be performed by the PI. Data handling and protection are conducted according to the ISO 14155 guidelines and ICH-GCP and applicable regulations.

677678679

The eCRF collects data from each participant. Specifically all data on each patient participating in the study are documented in the eCRF. The eCRF contains data items as specified in this CIP. Modification of the eCRF will be made only if deemed necessary and in accordance with any amendment to the CIP.

681 682

680

The patient's hospital records are stored securely in the hospital's EHR (Epic Systems Corporation, Verona, Wisconsin, USA).



Non-operative treatment of pediatric lateral humeral condyle fractures


| 716 | 18.1 Final Study Report |
|---|---|
| 715 | 18 Study report and publication policy |
| 714 | Patient Compensation Association (Patienterstatningen). |
| 713 | As with any treatment in the Danish healthcare system all patients are insured and covered by The |
| 712 | 17 Patient insurance |
| 711 | All expenses are paid for by the sponsor. |
| 710 | |
| 709 | Participants do not receive any economic benefits or gifts from the participation in this project. |
| 708 | |
| 707 | related to the subject of this project. The investigators declare that they have no conflict of interest. |
| 705<br>706 | The initiative for this study has been taken solely by the investigators. The investigators and affiliated colleagues have not received any financial payments or other benefits from any commercial entity |
| 704 | 16 Disclosures and economy |
| 703 | study progress and events according to their specific regulations and procedures. |
| 702 | be sent to a respective EC for evaluation and approval. The relevant EC will be kept informed about the |
| 701 | The CIP, associated documents, investigator's financial disclosure, the patient information and ICFs will |
| 700 | 15 Regulatory affairs |
| 699 | and approval for the access. |
| 698 | informed consent document will contain information about the confidentiality of the medical information |
| 697 | carried out by the PI. Personal medical information will be treated as confidential at all times. The |
| 696 | Fully identifiable information may be reviewed for the purpose of verifying data in the eCRF. This can be |
| 695 | i mady and confidentiality of the patient's medical data will be maintained through the study. |
| 693<br>694 | <b>14.3 Confidentiality</b> Privacy and confidentiality of the patient's medical data will be maintained through the study. |
| 692 | system (PACS). |
| 691 | Radiographs and MRIs are stored securely in the hospital's Picture archiving and communication |
| 690 | 14.2 Imaging data |
| 689 | after a patient's visit (i.e. 14 days after occurrence of a documentable event). |
| 688 | Data Capture (RedCAP, Vanderbilt University, USA). The eCRF is to be completed in a timely manner |
| 687 | to the eCRF is password protected. The project's eCRF is stored securely using Research Electronic |
| 685<br>686 | <b>14.1.1 Electronic CRF</b> For this study, an eCRF is designed to accommodate the specific features of the study design. Access |
| 005 | 14.1.1 Floatronic CDF |

The results of the statistical evaluation will be summarized in a report, which forms the basis for the

comprehensive FSR. The comprehensive FSR forms the basis for all future publications.

717



18.2 Publication

719

754755756

Non-operative treatment of pediatric lateral humeral condyle fractures


| 720<br>721 | The study protocol and the trial will be registered with Clinicaltrials.gov |
|---|---|
| 722 | The results, both positive, negative and inconclusive, will be sent for submission in a peer reviewed |
| 723 | international orthopedic journal, and the results will be presented at national and international scientific |
| 724 | meetings. Reporting will adhere to the STROBE guidelines for cohort studies [31]. |
| 725 | 19 Termination criteria |
| 726 | The progress of the study, in particular the enrollment and safety aspects, will be closely monitored |
| 727 | together with the sponsor. The sponsor may decide to terminate the. In case of an early study |
| 728 | termination, all patients already enrolled in the study will be followed up until the last FU visit as defined |
| 729 | in the CIP. |
| 730 | 19.1 Stopping rules |
| 731 | The recruitment will be put on hold for safety reason if: |
| 732 | |
| 733 | <ul> <li>Secondary displacement of more than 2 mm during FU in &gt; 75% of cases at interim analysis.</li> </ul> |
| 734 | The control of the control of the Control of the Co |
| 735<br>736 | In such a case, the reported complication will be discussed with the sponsor. The sponsor will decide about the actions to be taken and if the study needs to be stopped or not. |
| 737 | 20 Deviations from the Clinical Investigation Plan |
| 738 | Deviations from the procedures as described in this CIP or altering the CIP without following a defined |
| 739 | process are not permitted. |
| 740 | |
| 741 | A CIP deviation is any non-adherence to the protocol that does not involve the inclusion/exclusion |
| 742 | criteria, primary efficacy variable, and GCP guidelines. CIP deviations are minor and do not impact the |
| 743 | study in a major way. CIP deviations are to be reported to the sponsor within ten working days. |
| 744 | |
| 745 | A CIP violation is any significant divergence from the protocol on the part of the patient, investigator, |
| 746 | sponsor, or any other responsible party that affects e.g. the inclusion/exclusion criteria, primary efficacy |
| 747 | variable, or GCP guidelines. Violations will be recorded at the study site and in the eCRF. |
| 748 | 21 Amendments to the Clinical Investigation Plan |
| 749 | No changes to the approved CIP are allowed, except when the change removes immediate threats for |
| 750 | the patient safety or is of a purely administrative or logistic nature. |
| 751 | |
| 752 | Should there be any need during the performance of the study to change this CIP, an amendment will |
| 753 | be developed, issued and approved by or notified to the required bodies. |




# 757 22 Time schedule

| Ethics Committee approvals | 28.06.2021 | to | 01.09.2021 |
|----------------------------|------------|----|------------|
| First patient/first visit | 01.10.2021 | | |
| Last patient/first visit | 01.10.2023 | | |
| Last patient/last visit | 01.10.2025 | | |
| Data analysis | 01.11.2025 | to | 01.03.2026 |
| Final Study Report | 01.03.2026 | to | 01.06.2026 |

### 23 Authors

### CIP developed by

759760

758

| PCI | Department of Orthopedic Surgery<br>Copenhagen University Hospital - Herlev<br>and Gentofte, Copenhagen, Denmark |
|---|---|
| Project Manager | Morten Jon Andersen |
| Additional author(s) | Peter Søndergaard, MD<br>Bo Sanderhoff Olsen, MD, ph.d., professor<br>Jeppe Vejlgaard Rasmussen, MD, ph.d. |

761 762

### CIP approval signatures

763 764

| Name | Function | Date | Signature |
|---|---|---|---|
| Morten Jon<br>Andersen | Principal Coordinating<br>Investigator | | |

765

| Name | Function | Date | Signature |
|------------------------|-------------------------|------|-----------|
| Bo Sanderhoff<br>Olsen | Director of institution | | |

766 767

768

769

770

771

772

773

774

775

776

777

778

With signing this statement, I agree and confirm:

- To have read and understood this CIP and to have informed and to have supervised the appropriate training of all research team members of this study site involved with the conduct of the study.
- To assume responsibility to conduct the study in compliance with this protocol and future amendments at this study site.
- To obtain written approval the independent EC before initiating the clinical investigation at this study site.
- To not implement any changes to the protocol or the corresponding procedures without written
  agreement from the sponsor and the EC, except where necessary to eliminate immediate risk to the
  study patients.
- That I and all team members involved in the conduct of this clinical investigation are aware and trained in aspects of ICH-GCP and all applicable regulatory requirements.





#### 24 Reference list

- 780 1. Rang M, Pring ME, Wenger DR. Rang's Children's Fractures. 3. udg. Lippincott Williams & Wilkins; 2005.
- Kamegaya M, Shinohara Y, Kurokawa M, et al. Assessment of stability in children's minimally displaced lateral humeral condyle fracture by magnetic resonance imaging. J Pediatr Orthop 1999;19:570–2.
- Horn BD, Herman MJ, Crisci K, et al. Assessment of stability in children's minimally displaced lateral humeral condyle fracture by magnetic resonance imaging. J Pediatr Orthop 2020;90:30–5.
- Horn BD, Herman MJ, Crisci K, et al. Fractures of the lateral humeral condyle: Role of the cartilage hinge in fracture stability. J Pediatr Orthop 2002;22:8–11.
- 5. Beltran J, Rosenberg ZS, Kawelblum M, et al. Pediatric elbow fractures: MRI evaluation. Skelet Radiol A J Radiol Pathol Orthop 1994;23:277–81.
- Houshian S, Mehdi B, Larsen MS. The epidemiology of elbow fracture in children: Analysis of 355 fractures, with special reference to supracondylar humerus fractures. J Orthop Sci 2001;
- 794 7. Waters PM, Skaggs DL, Flynn JM (Jack), et al. Rockwood and Wilkins' fractures in children. 9. udg. Wolters Kluwer; 2019.
- Naranje SM, Erali RA, Warner WC, et al. Epidemiology of Pediatric Fractures Presenting to Emergency Departments in the United States. J Pediatr Orthop 2016;36:e45–8.
- Hedström EM, Svensson O, Bergström U, et al. Epidemiology of fractures in children and
   adolescents: Increased incidence over the past decade: A population-based study from northern
   Sweden. Acta Orthop 2010;81:148–53.
- Rennie L, Court-Brown CM, Mok JYQ, et al. The epidemiology of fractures in children. Injury 2007;38:913–22.
- Landin LA, Danielsson LG. Elbow fractures in children: An epidemiological analysis of 589 cases. Acta Orthop 1986;57:309–12.
- Pirker ME, Weinberg AM, Höllwarth ME, et al. Subsequent displacement of initially nondisplaced and minimally displaced fractures of the lateral humeral condyle in children. J Trauma Inj Infect Crit Care 2005;58:1202–7.
- Abzug JM, Dua K, Kozin SH, et al. Current Concepts in the Treatment of Lateral Condyle Fractures in Children. J Am Acad Orthop Surg 2019;00:1.
- Song KS, Kang CH, Min BW, et al. Internal oblique radiographs for diagnosis of nondisplaced or minimally displaced lateral condylar fractures of the humerus in children. J Bone Jt Surg Ser A 2007;89:58–63.
- Goodwin SJ, Irwin LJ, Irwin GJ. Gender differences in the order of appearance of elbow ossification centres. Scott Med J 2019;64:2–9.
- Shrader W, Campbell M, Jacofsky D. Accuracy of emergency room physicians' interpretation of elbow fractures in children. Orthopedics Orthopedics; 2008;31:1177.
- Milch H. Fractures and fracture dislocations of the humeral condyles. J Trauma Inj Infect Crit Care 1964;4:592–607.
- Song KS, Chul HCK, Byung WM, et al. Closed reduction and internal fixation of displaced unstable lateral condylar fractures of the humerus in children. J Bone Jt Surg Ser A 2008;90:2673–81.







- Bast SC, Hoffer MM, Aval S. Nonoperative treatment for minimally and nondisplaced lateral humeral condyle fractures in children. J Pediatr Orthop 1998;18:448–50.
- Weiss JM, Graves S, Yang S, et al. A new classification system predictive of complications in surgically treated pediatric humeral lateral condyle fractures. J Pediatr Orthop 2009;29:602–5.
- Haillotte G, Bachy M, Delpont M, et al. The Use of Magnetic Resonance Imaging in Management of Minimally Displaced or Nondisplaced Lateral Humeral Condyle Fractures in Children. Pediatr Emerg Care 2017;33:21–5.
- Thévenin-Lemoine C, Salanne S, Pham T, et al. Relevance of MRI for management of nondisplaced lateral humeral condyle fractures in children. Orthop Traumatol Surg Res 2017;103:777–81.
- Runge SB, Christensen NL, Jensen K, et al. Children centered care: Minimizing the need for anesthesia with a multi-faceted concept for MRI in children aged 4–6. Eur J Radiol Elsevier; 2018;107:183–7.
- Hallowell LM, Stewart SE, De Amorim E Silva CT, et al. Reviewing the process of preparing children for MRI. Pediatr Radiol Pediatr Radiol; 2008. s. 271–9.
- Raschle NM, Lee M, Buechler R, et al. Making MR imaging child's play Pediatric neuroimaging protocol, guidelines and procedure. J Vis Exp 2009;29:1–6.
- De Bie HMA, Boersma M, Wattjes MP, et al. Preparing children with a mock scanner training protocol results in high quality structural and functional MRI scans. Eur J Pediatr 2010;169:1079–85.
- Cahoon GD, Davison TE. Prediction of compliance with MRI procedures among children of ages 3 years to 12 years. Pediatr Radiol 2014;44:1302–9.
- Ahmad R, Hu HH, Krishnamurthy R, et al. Reducing sedation for pediatric body MRI using accelerated and abbreviated imaging protocols. Pediatr Radiol Pediatr Radiol; 2018;48:37–49.
- Barnea-Goraly N, Weinzimer SA, Ruedy KJ, et al. High success rates of sedation-free brain MRI scanning in young children using simple subject preparation protocols with and without a commercial mock scanner-the Diabetes Research in Children Network (DirecNet) experience.

  Pediatr Radiol 2014;44:181–6.
- Vandenbroucke JP, Von Elm E, Altman DG, et al. Strengthening the Reporting of Observational Studies in Epidemiology (STROBE): Explanation and elaboration. Epidemiology 2007;18:805–35.
- Dill T. Contraindications to magnetic resonance imaging: non-invasive imaging. Heart England; 2008;94:943–8.
- Tawfik AI, Kamr WH, Taman SE. Comparison of 2D Fat Suppressed Proton Density (FS-PD) and 3D (WATS-c) MRI pulse sequences in evaluation of chondromalacia patellae. Egypt J Radiol Nucl Med 2019;50:85.
- Bitar R, Leung G, Perng R, et al. MR pulse sequences: What every radiologist wants to know but is afraid to ask. Radiographics 2006. s. 513–37.
- 35. Morrey BF. The elbow and its disorders. Saunders; 2008.
- 863 36. Longo UG, Franceschi F, Loppini M, et al. Rating systems for evaluation of the elbow. Br Med Bull 2008;
- 865 37. Cusick MC, Bonnaig NS, Azar FM, et al. Accuracy and reliability of the mayo elbow performance



866

score. J Hand Surg Am 2014;

Non-operative treatment of pediatric lateral humeral condyle fractures


| 867<br>868 | 38. | Merkel, Voepel-Lewis, Shayevitz, et al. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs 1997;23:293–7. |
|---|---|---|
| 869<br>870 | 39. | Hicks CL, Von Baeyer CL, Spafford PA, et al. The Faces Pain Scale - Revised: Toward a common metric in pediatric pain measurement. Pain 2001;31:1177. |
| 871<br>872<br>873 | 40. | Bieri D, Reeve RA, Champion GD, et al. The faces pain scale for the self-assessment of the severity of pain experienced by children: Development, initial validation, and preliminary investigation for ratio scale properties. Pain 1990;41:139–50. |
| 874<br>875 | 41. | Huguet A, Stinson JN, McGrath PJ. Measurement of self-reported pain intensity in children and adolescents. J Psychosom Res 2010;68:329–36. |
| 876<br>877 | 42. | Bailey B, Gravel J, Daoust R. Reliability of the visual analog scale in children with acute pain in the emergency department. Pain 2012;153:839–42. |
| 878 | | |



879

# **Appendix 1 - Diagnosis and Treatment Protocol**

